CLINICAL TRIAL: NCT00068133
Title: A Phase II Multicenter, Double-Blind, Placebo-Controlled, Trial of VLTS-589 in Subjects With Intermittent Claudication Secondary to Peripheral Arterial Disease
Brief Title: Trial of VLTS-589 in Subjects With Intermittent Claudication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valentis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VLTS-589-121
Record Dates: First submitted 2003-09-08; First posted 2003-09-10 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases

INTERVENTIONS:
Genetic: Plasmid based Gene Transfer product-VLTS-589

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of VLTS-589 compared with placebo, administered bilaterally to the lower extremities, in subjects with intermittent claudication and to determine the effect of VLTS-589 in peak walking time (PWT) for subjects receiving VLTS-589 compared with subjects receiving placebo.

ELIGIBILITY:
Inclusion criteria:

* Men or women between 40 and 80 years of age,
* Must give informed consent,
* Current medical history of peripheral arterial disease, which includes the following symptoms: leg pain, leg discomfort or leg weakness

Exclusion criteria:

* Ulcers or gangrene,
* History of cancer (except skin cancer) within the past 5 years,
* Participation in another clinical trial within 30 days of enrollment in this trial,
* Unwillingness or inability to comply with all study requirements

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Cardiology Pc, Birmingham, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Access Clinical Trials-Cardiovascular Research, Beverly Hills, California
  - Jacksonville Heart Center, Jacksonville, Florida
  - Heart Specialists of Sarasota Clinical Research Center, Sarasota, Florida
  - American Cardiovascular Research Institute, Atlanta, Georgia
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Prairie Heart Institution at St. John's Hospital, Springfield, Illinois
  - The Care Group, Indianapolis, Indiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Minneapolis Heart Institution Foundation, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - St. Vincent's Hospital, New York, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Methodist Hospital, Houston, Texas
  - Daniel Gottleib, MD, Seattle, Washington